CLINICAL TRIAL: NCT01050153
Title: An Evaluation of the Clinical Utility of Thrombelastography (TEG) in Guiding Low Molecular Weight Heparin (LMWH) and Antiplatelet Prophylaxis of Venous Thromboembolism (VTE) Following Trauma
Brief Title: The Clinical Utility of Thrombelastography in Guiding Prophylaxis of Venous Thromboembolism Following Trauma
Acronym: VTEPX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Ernest E. Moore, MD, Chief, Department of Surgery and Trauma Services Rocky Mountain Regional Trauma Center, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COMIRB # 09-0753
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Venous Thromboembolism
Keywords: Prevention of venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dalteparin; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (standard of care) (Active Comparator): Dalteparin sodium 5000IU subcutaneously daily
  Interventions: Drug: Dalteparin sodium
- TEG-guided thromboprophylaxis (Experimental): Dalteparin sodium plus/minus anti-platelet medication (aspirin) per a TEG-guided algorithm
  Interventions: Drug: Dalteparin sodium/aspirin

INTERVENTIONS:
Drug: Dalteparin sodium — Dalteparin sodium injection 5000IU subcutaneously daily until fully ambulatory
  Other Names: Dalteparin sodium (Fragmin)
  Arms: Control (standard of care)
Drug: Dalteparin sodium/aspirin — Dalteparin sodium (2500-10,000IU sc daily), aspirin (81-325mg daily) po.
  Other Names: dalteparin sodium (Fragmin)
  Arms: TEG-guided thromboprophylaxis

SUMMARY:
This study plans to learn more about how to prevent blood clots in the veins of your extremities. You are at risk of forming these clots after a major injury and when you have had surgery and are hospitalized on bed rest.

Usually, patients in the SICU at Denver Health who are at risk for blood clots receive preventative treatment with a FDA-approved medicine called Fragmin. Fragmin is intended to prevent blood clots from forming but, with the way it is generally used, some patients may still develop blood clots. All patients treated with Fragmin to prevent blood clots at Denver Health, currently receive the same Fragmin dose. This treatment is called the "standard of care".

So far, in the US, there has not been a commonly available test that can tell us:

* if the standard dose of Fragmin is enough to prevent blood clots for everyone, or
* if different patients need different doses, or
* if other blood clot preventing medicines, that work in a different way, should be used in addition to Fragmin.

The ability of your blood to clot and the strength of the clot formed can be described by a FDA-approved blood test called thrombelastography, referred to as TEG. TEG may provide us with answers to each of the questions above. Our preliminary data indicate that it is helpful in assessing both clotting and bleeding tendencies and may prove useful in guiding treatment for the prevention of blood clots.

The aim of this study is to determine if a treatment plan using Fragmin, and, if indicated, one or two additional FDA-approved medicines called anti-platelet drugs, guided by the results of TEG testing, may be better at preventing blood clots than our current standard of care.

DETAILED DESCRIPTION:
This preliminary/pilot study involves a prospective, randomized, open-label, parallel group comparison of Denver Health's current standard of care for prevention of venous thromboembolism (VTE), commonly known as blood clots, using LMWH (Fragmin) 5000IU subcutaneously daily, with a thrombelastography (TEG)-guided, algorithm-based, individualized regimen of LMWH (Fragmin) plus/minus anti-platelet therapy (aspirin) guided by platelet mapping, in patients admitted to the SICU following trauma.

Approximately 50 trauma patients for whom prevention of VTE with LMWH is indicated, will be enrolled over a six month period.

The specific aims of this study are as follows:

1. To determine the incidence of, and to characterize, hypercoagulability using TEG and conventional clinical coagulation testing (APTT, INR), Antithrombin III levels and Protein C activity.
2. In the group of patients receiving LMWH (Fragmin) therapy alone for prevention of VTE:

   1. to assess the anticoagulant effect of standard LMWH (Fragmin) dosing (5000IU subcutaneously once daily) using TEG and Anti-Factor Xa level measurement, and
   2. to determine the extent of correlation of relevant TEG parameters with measured Anti-Factor Xa levels (U/ml).
3. To assess whether TEG is a useful clinical tool for monitoring and optimizing prophylactic LMWH (Fragmin) therapy and for identifying the need for anti-platelet therapy to minimize the risk of VTE in these patients.
4. To evaluate the clinical utility of platelet mapping for guiding anti-platelet therapy in those patients for whom it is indicated by TEG results.
5. To determine the incidence of deep vein thrombosis (DVT) and pulmonary embolism (PE) in each randomized group and in the subgroup receiving anti-platelet therapy in addition to LMWH (Fragmin) for prevention of VTE.

The overall aim is to utilize the above data to evaluate a) the adequacy of our standard Fragmin dosing regimen (5000IU subcutaneously once daily) alone for prevention of VTE in our trauma/SICU patients, b) the need for anti-platelet agents in addition to LMWH (Fragmin) for prevention of VTE in our population, and c) to validate/further develop the TEG-guided algorithm for optimal prophylaxis of VTE using LMWH (Fragmin) plus/minus anti-platelet therapy guided by platelet mapping.

ELIGIBILITY:
Inclusion Criteria:

* age at least 18 years,
* blunt or penetrating trauma requiring admission to the SICU
* requirement for LMWH (Fragmin) therapy for prophylaxis of VTE as standard of care, and
* informed consent by patient, legally authorized representative or proxy decision maker (if patient incompetent to provide) obtained and documented.

Exclusion Criteria:

Presence of any of the following absolute contraindications to LMWH (Fragmin) therapy:

* known hypersensitivity to dalteparin sodium,
* known hypersensitivity to heparin or pork products,
* thrombocytopenia associated with positive tests for antiplatelet antibody in the presence of Fragmin,
* history of heparin-induced thrombocytopenia (HIT),
* chronic liver disease (bilirubin >2 mg/dl) or kidney insufficiency (CrCl <30mL/min),
* intravascular thrombolytic therapy within 24 hours,
* resuscitation that required massive transfusion (>10 units RBC within 6 hours),
* ongoing resuscitation for hemorrhagic shock,
* known bleeding disorder or coagulopathy (INR >2 not on warfarin),
* thrombocytopenia (platelets <20K/uL),
* subdural or epidural hematoma.

Or

Presence of any of the following relative contraindications to LMWH (Fragmin) therapy:

* new intracranial lesions, neoplasms or monitoring devices,
* extravascular thrombolytic therapy,
* severe uncontrolled hypertension,
* arterial dissection
* recent (within 12 hours) intraocular surgery (prior or planned),
* recent (within 72 hours) intracranial or spine surgery (prior or planned),
* conditions associated with increased risk of hemorrhage, e.g. active gastrointestinal ulceration, angiodysplastic disease, gastrointestinal bleeding within the past six months, bacterial endocarditis, history of hemorrhagic stroke, diabetic retinopathy.

Or

Presence, or removal within the last 12 hours, of an indwelling epidural or spinal catheter, OR recent (within the last 12 hours) or planned neuraxial (spinal/epidural) anesthesia or spinal puncture.

Or

Per history taken from patient or family, concomitant or known use within one week prior to hospitalization, of drugs affecting hemostasis such as NSAIDS, platelet inhibitors or other anticoagulants, except as specified in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest E. Moore Jr, M.D., Principal Investigator — Chief, Department of Surgery and Trauma Services , Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

REFERENCES:
- See also: Related Info — http://denverhealth.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 consecutive eligible patients admitted to the Surgical Intensive Care Unit following trauma between March 2010 and December 2011 were enrolled in the study.
Groups:
- Control (Standard of Care): Dalteparin sodium 5000IU subcutaneously daily
  Dalteparin sodium : Dalteparin sodium injection 5000IU subcutaneously daily until fully ambulatory
- TEG-guided Thromboprophylaxis: Dalteparin sodium plus/minus anti-platelet medication (aspirin) per a TEG-guided algorithm
  Dalteparin sodium/aspirin : Dalteparin sodium (2500-10,000IU sc daily), aspirin (81-325mg daily)po.
Period: Overall Study
Arm/Group | Control (Standard of Care) | TEG-guided Thromboprophylaxis
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Standard of Care) | TEG-guided Thromboprophylaxis | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.04 (12.18) | 38.44 (14.34) | 39.24 (13.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 19 | 17 | 36
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Hypercoagulability
Description: To determine the incidence of, and to characterize, hypercoagulability in a sample of trauma patients admitted to the SICU at DHMC using TEG and conventional clinical coagulation testing (APTT, INR), antithrombin III levels and protein C activity. Hypercoagulability is defined as TEG parameter G (clot strength) >10.9.
Time Frame: Study day five.
Population: The reason for having 21 participants in the Control group and 18 participants in the TEG-guided group is that 21 and 18 participants in the respective groups stayed five days or longer. Four participants (25-21) in the Control group and seven participants (25-18) in the TEG-guided group stayed less than five days.
Measure: Number; unit: participants
Arm/Group | Control (Standard of Care) | TEG-guided Thromboprophylaxis
Number analyzed (Participants) | 21 | 18
participants | 16 | 18

2. Primary Outcome: Incidence of VTE
Description: The incidence and nature of hypercoagulability and the incidence of deep vein thrombosis and pulmonary embolism in each randomized group and in the subgroup receiving anti-platelet therapy in addition to Fragmin (descriptive analysis only)
Time Frame: Day 28 or discharge, whichever comes first.
Measure: Number; unit: participants
Arm/Group | Control (Standard of Care) | TEG-guided Thromboprophylaxis
Number analyzed (Participants) | 25 | 25
participants | 0 | 0

3. Secondary Outcome: TEG Parameters
Description: R is a reaction time. The time from the start of a sample run until the first significant levels of detectable clot formation (amplitude = 2 mm in the TEG tracing).
  Rf is a difference in reaction time between Fragmin-active and Fragmin-neutralized samples.
  Achievement of a certain clot strength K is a measure of the time from R until a fixed level of clot strength is reached (amplitude = 20 mm).
  Angle or α measures the rapidity of fibrin build-up and cross-linking (clot strengthening). This most represents fibrinogen level. Angle relates to K, since both are a function of the rate of clot formation.
  MA, or Maximum Amplitude, is a direct function of the maximum clot strength. In tests where platelets are part of the clot, this parameter most reflects platelet function/aggregation. Clot strength is the result of two components - the modest contribution of fibrin and the much more significant contribution of the platelets.
Time Frame: Study day five.
Measure: Mean (Standard Error); unit: Minutes
Arm/Group | Control (Standard of Care) | TEG-guided Thromboprophylaxis
Number analyzed (Participants) | 21 | 18
Minutes
  R value | 5.89 (0.38) | 5.83 (0.35)
  Rf value | -0.09 (0.09) | -0.34 (0.16)

4. Secondary Outcome: International Normalized Ratio (INR)
Description: Plasma based conventional coagulation testing parameters
Time Frame: Study day five.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Control (Standard of Care) | TEG-guided Thromboprophylaxis
Number analyzed (Participants) | 20 | 19
ratio | 1.23 (0.19) | 1.13 (0.09)

5. Secondary Outcome: Platelet Count
Description: Platelet count measured by CBC test
Time Frame: Study day five.
Measure: Mean (Standard Deviation); unit: * 10^3 platelets/µL
Arm/Group | Control (Standard of Care) | TEG-guided Thromboprophylaxis
Number analyzed (Participants) | 22 | 21
* 10^3 platelets/µL | 261.64 (171.73) | 267.76 (83.23)

6. Secondary Outcome: TEG Parameters
Description: Shear elastic modulus strength (SEMS). The MA parameter can be transformed into the actual measure of clot strength (G) using the formula below, and is measured in dyn/cm2 divided by 1000 (displayed in the software as Kd/sc).
  The absolute SEMS of the sample can be calculated from MA as follows:
  G = (5000MA/(100-MA))/1000 An amplitude of 50 mm corresponds to a SEMS of 5000 dyn/cm2. An increase in MA from 50 mm to 67 mm is equivalent to a two-fold increase in the SEMS. The G parameter not only provides a measurement of clot firmness in force units, but also is more indicative of small changes in the clot strength or clot breakdown than is the amplitude in mm because it is an exponential reflection of MA.
Time Frame: Study day five.
Measure: Mean (Standard Error); unit: Kd/sc
Arm/Group | Control (Standard of Care) | TEG-guided Thromboprophylaxis
Number analyzed (Participants) | 21 | 18
Kd/sc | 14.97 (0.91) | 15.46 (0.60)

7. Secondary Outcome: Conventional Coagulation Testing Parameters
Description: Plasma based conventional coagulation testing parameters - Anti Xa
Time Frame: Study day five.
Measure: Mean (Standard Error); unit: IU/mL
Arm/Group | Control (Standard of Care) | TEG-guided Thromboprophylaxis
Number analyzed (Participants) | 20 | 19
IU/mL | 0.14 (0.01) | 0.18 (0.01)

8. Secondary Outcome: Conventional Coagulation Testing Parameters
Description: Plasma based conventional coagulation testing parameters - Fibrinogen
Time Frame: Study day five.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Control (Standard of Care) | TEG-guided Thromboprophylaxis
Number analyzed (Participants) | 20 | 19
mg/dL | 691.4 (146.69) | 687.11 (157.75)

9. Secondary Outcome: Conventional Coagulation Testing Parameters
Description: Plasma based conventional coagulation testing parameters - Anti-thrombin III
Time Frame: Study day five.
Measure: Mean (Standard Error); unit: percentage of activity
Arm/Group | Control (Standard of Care) | TEG-guided Thromboprophylaxis
Number analyzed (Participants) | 20 | 19
percentage of activity | 79.3 (4.31) | 80 (4.31)

10. Secondary Outcome: Conventional Coagulation Testing Parameters
Description: Plasma based conventional coagulation testing parameters - Protein C
Time Frame: Study day five.
Measure: Mean (Standard Error); unit: percentage of activity
Arm/Group | Control (Standard of Care) | TEG-guided Thromboprophylaxis
Number analyzed (Participants) | 20 | 19
percentage of activity | 76.65 (6.17) | 79.83 (7.6)

ADVERSE EVENTS:
Arm/Group | Control (Standard of Care) | TEG-guided Thromboprophylaxis
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 1/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (Standard of Care) (N=25) | TEG-guided Thromboprophylaxis (N=25)
Decrease in Hemoglobin level more than 2g/dL in 24 hour period. (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
1. lower than expected incidence of VTE events
2. Control group patients were followed for 5 days, while TEG-guided group was followed as long as in SICU
3. adherence to VTE prophylaxis with Daltaparin was significantly low in the TEG-guided group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No